CLINICAL TRIAL: NCT07160205
Title: A Phase 2-Phase 3, Double-blinded, Randomized, Dose-repeating, Cross-over Study to Assess the Safety and Efficacy of Allogeneic ULSC on Disease Severity and Steroid Tapering in Participants With Dermatomyositis/ Polymyositis (DM/PM)
Brief Title: Safety and Efficacy of ULSC on Disease Severity and Steroid Tapering in Participants With Dermatomyositis/ Polymyositis (DM/PM), Also Known as Idiopathic Inflammatory Myopathy (IIM)
Acronym: IIMPACT
Status: Recruiting | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Restem, LLC. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Treatment
Other Study IDs: RES001-DMPM-02
Record Dates: First submitted 2025-08-26; First posted 2025-09-08 (Actual); Last update posted 2026-02-03 (Actual); Status verified 2026-01

CONDITIONS: Idiopathic Inflammatory Myositis (IIM); DERMATOMYOSITIS OR POLYMYOSITIS
MeSH Terms: conditions — Myositis; Dermatomyositis

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Cohort 1: ULSC first; Placebo second (Experimental): Cohort 1 will receive 1.5 x 10^8 ULSC per dose through IV infusion on Day 0, Month 3, and Month 6 (total of three doses). One month after the third dose, Cohort 1 will cross-over to receive Placebo IV infusion on Month 7, Month 10, and Month 13.
  Interventions: Biological: ULSC (1.5 x 10^8 cells/dose); Biological: Placebo (no cells)
- Cohort 2: Placebo first; ULSC second (Experimental): Cohort 2 will receive Placebo IV infusion on Day 0, Month 3, and Month 6 (total of three Placebo infusions). One month after the third dose, Cohort 2 will cross-over to receive 1.5 x 10^8 ULSC per dose through IV infusion on Month 7, Month 10, and Month 13.
  Interventions: Biological: ULSC (1.5 x 10^8 cells/dose); Biological: Placebo (no cells)

INTERVENTIONS:
Biological: ULSC (1.5 x 10^8 cells/dose) — Allogeneic umbilical-cord lining stem cells (ULSC) are cryopreserved and supplied in vials to be thawed and prepared for infusion at point of use. Each dose of 1.5 x 10^8 ULSC will be added into 250 sterile saline IV bag for infusion (total volume of 260 mL volume).
Biological: Placebo (no cells) — The Placebo will be 250 ml sterile saline with vehicle (total volume of 260 mL) IV bag for infusion.

SUMMARY:
The goal of this clinical trial is to learn about how an umbilical cord lining-derived stem cell (ULSC) product performs when treating Dermatomyositis/Polymyositis (DM/PM), also known as idiopathic inflammatory myopathy (IIM) in adults. It will assess safety and efficacy in relieving symptoms of DM/PM with ULSC administered in three intravenous (IV) doses of 150 million cells per dose.

The main questions that this study plans to answer are:

* Is ULSC as safe as placebo (a look-alike saline without cells) in repeated IV infusion?
* Does ULSC improve symptoms of DM/PM after three doses? Researchers will compare ULSC to placebo and evaluate changes from baseline (before first dose) to after each dose and after all three doses are completed per treatment study period.
* For participants undergoing steroid (e.g., prednisone) therapy for DM/PM, does ULSC allow their steroid dose to be reduced? Does ULSC reduce need for rescue therapy?

Participants will have been diagnosed with either DM or PM:

* Diagnosed according to the EULAR/ACR 2017 Classification Criteria for idiopathic inflammatory myositis (IIM), which includes DM and PM.
* Positive for myositis-associated antibody or undergone evaluation to exclude mimics.

Participants in this study will:

* Participate for total of 25 months with 15 in-person clinic visits and 8 virtual visits on phone or video call.
* Receive both ULSC and placebo for a total of 6 IV infusions (260 mL) 3 months apart.
* Receive 3 doses of ULSC and 3 doses placebo in either of two sequences, as assigned: ULSC first and placebo second, or placebo first and ULSC second.
* If undergoing steroid therapy, will have steroid dose taper prescribing lower doses starting two weeks after the second infusion.
* Return for follow-up visits after each dose and up to 12 months after final dose.
* Have follow-ups including self-reported questionnaires, physical exam, muscle strength and endurance tests, blood tests, pulmonary function tests, and other assessments.

ELIGIBILITY:
Inclusion Criteria:

1. Participants will be ≥18 years old.
2. Diagnosis of idiopathic inflammatory myositis (IIM) based on 2017 EULAR/ACR Classification Criteria for adult IIM, corresponding to a score of ≥ 5.5 (≥ 6.7 with muscle biopsy).
3. Active disease as defined by any one of the following test results:

   1. Elevated Creatine Kinase (CK) or Aldolase (more than 1.5 x the upper limit of normal) at screening, OR
   2. MRI positive for active, muscle inflammation within 12 weeks prior to screening, OR
   3. EMG read as active myositis within 12 weeks prior to screening, OR
   4. muscle biopsy obtained within 12 weeks of the screening showing active inflammatory disease.
4. Muscle weakness or active cutaneous manifestations of dermatomyositis assessed at Screening and documented with either of the following scores:

   1. Bilateral MMT-8 score of ≤142/150, OR
   2. CDASI Total Activity score of ≥ 7.
5. Participants must be receiving standard of care treatment with one or more immunosuppressants or at least 5 mg prednisone (or corticosteroid equivalent).

   1. Immunosuppressive doses should be stable for at least 12 weeks prior to enrollment. Participants must remain on stable immunosuppressive therapy for the duration of the trial unless discontinuation is warranted due to toxicity or another clinical reason.
   2. Hydroxychloroquine (HCQ) doses should be stable for at least 12 weeks prior to enrollment.
   3. Steroid doses should be stable for at least 4 weeks prior to enrollment. At screening and enrollment, maximum dose allowed is 25 mg/day prednisone (or corticosteroid equivalent).
   4. Allowed immunosuppressants include: methotrexate, azathioprine, mycophenolate, cyclosporine, IVIG, and others to be evaluated at the discretion of the investigator.
6. Participants will either be:

   1. positive for a myositis-associated antibody, OR
   2. will have undergone evaluation to exclude mimics, as deemed appropriate by the Investigator.

   Note: The minimum workup to be performed on all prospective participants to exclude mimics is as standardly followed, which may include:
   * Medical history and physical exam to determine the clinical course and progression of symptoms, the distribution of weakness, and the absence of features of myelopathy, neuropathy, neuromuscular disease, myotonic dystrophy, and congenital myopathy;
   * Elevated Creatine Kinase (CK) or Aldolase levels in blood;
   * Electromyography (EMG) and/or MRI of clinically affected 99+proximal muscle group;
   * Myositis-specific and myositis-associated autoantibodies in blood;
   * Muscle biopsy with characteristic features of IIM and excluding features of muscular dystrophy, metabolic myopathies, drug-induce myopathy, inclusion body myopathy, and necrotizing myopathy;
   * Blood tests for exclusion of HIV, Hepatitis B (HBV), and Hepatitis C (HCV). [Screening tests are done for HIV ELISA, HBs Ag, HBc Ab, and HCV Ab with reflex for HCV RNA (PCR) for exclusion criteria.]
7. Adequate pulmonary function, defined as saturated oxygen (SpO2 ≥ 94%) on room air.
8. Left ventricular ejection fraction (LVEF) ≥ 30% as assessed by echocardiogram (ECHO) or multigated acquisition (MUGA) scan performed within 8 weeks prior to Screening.
9. Participants must have the ability to comply with the requirements of the study.
10. All participants of reproductive age/capacity will be required to use adequate contraception, defined as at least one form of a highly effective contraceptive (i.e., condoms, hormonal birth control, IUD), with any partners during the study period and for at least three months beyond the study period, for safety.
11. Participant will have the ability to understand and provide written informed consent.

Exclusion Criteria:

The presence of any of the following criteria excludes a participant from study enrollment:

1. A diagnosis of inclusion body myositis, juvenile DM or PM, myositis in the context of significant autoimmune rheumatologic disease.
2. Diagnosis of IIM as part of an overlap syndrome (except overlap with Sjogren's syndrome).
3. Initiation of Rituxan (rituximab) treatment within 12 weeks of randomization. If participant is already on Rituxan, they must remain on a stable dose throughout the trial.
4. Use of other biologic or investigational drug within 6 half-lives for the agent.
5. Diagnosis of myositis-associated interstitial lung disease or cardiac involvement sufficient to limit participation in the trial in the discretion of the PI.
6. End-stage IIM with irreversible muscle involvement seen on biopsy.
7. Patients with predominant muscle atrophy secondary to uncontrolled or chronic DM or PM, based on clinical, biochemical, and/or radiologic assessment, despite previous optimized treatment.
8. Non-immune myopathies.
9. Cancer associated with myositis.
10. Hypersensitivity to study product components including history of hypersensitivity to dimethyl sulfoxide (DMSO).
11. Pregnant or lactating participants.
12. Concomitant severe cardiac, pulmonary disease, active infection, or other conditions that preclude assessment of safety and efficacy of the study product.
13. Anticipated need for surgery during the trial period.
14. A history of prevalent noncompliance with medical therapy.
15. Recipient of an organ transplant.
16. Neutropenia [absolute neutrophil count <1,800/mm^3 (or <1,000/mm^3 in African-American participants)].
17. Severe impairment in renal function (estimated glomerular filtration rate <30 ml/kg*min).
18. Recent or planned use of vaccination with live attenuated viruses.
19. Active cancer or prior diagnosis of cancer within the past 2 years, except non-melanoma skin cancer and carcinoma in situ of cervix Potential participants diagnosed with IIM <3 years before screening will have mandatory evaluation for cancer.
20. Participants with current or prior hepatitis B infection that could be at risk for reactivation. [For eligibility, screening test results must be HBsAg (DNA) negative and anti-HBc (core antibody total) negative).]
21. Participant with HIV or active Hepatitis C. [For eligibility, the following screening tests must have negative or non-reactive results: HIV ELISA, HCV Ab with reflex for HCV RNA (PCR); if HCV Ab test is positive, exclude if HCV RNA (PCR) is positive.]
22. Condition that would impair an assessment of muscle strength, including neurological disorders such as Parkinson's disease or severe musculoskeletal condition.
23. Any other condition that, in the judgment of the Investigator or Sponsor, would be a contraindication to enrollment, study product administration, or follow-up.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2026-01-06 (Actual); Primary Completion 2028-09 (Estimated); Study Completion 2029-08 (Estimated)

PRIMARY OUTCOMES:
Safety based on Adverse Events (AEs) and Serious Adverse Events (SAEs) that begin during or following treatment infusion. | Each visit from Day 0, 7 days, and 30 days after each infusion, and all follow-up visits up to 12 months after the final treatment infusion.
  Cumulative listing of all AEs/SAEs per cohort with descriptive statistics for categorical variables and count variables to compare between ULSC and Placebo, with emphasis on All SAEs and AEs/SAEs suspected to be treatment infusion-related.
Efficacy based on Total Improvement Score (TIS, expressed as continuous variable) in the 2016 ACR/EULAR Myositis Response Criteria | From baseline (i.e., before first dose per treatment) to 7 months (i.e., one month after the third/final dose per treatment) for each treatment group and each study period.
  Total Improvement Score (TIS) as continuous variable (scale of 0 to 100 points) will be assessed; TIS is a weighted average of the sub-scores in the 6 core set measures that comprise the validated outcome measure in the 2016 ACR/EULAR Myositis Response Criteria.

SECONDARY OUTCOMES:
Need for Rescue Therapy (Incidence) | From baseline to 7 months for both study periods.
  The incidence of need for rescue therapy will be assessed by the number of participants that require administration of rescue therapy.
Need for Rescue Therapy (Time) | From baseline to 7 months for both study periods.
  Need for rescue therapy will be assessed in terms of the time to rescue therapy, i.e. time from the first dose of study treatment to the first administration of rescue therapy required.
Glucocorticoid Dose (prednisone equivalents per day) Tapering | From baseline to 4 months and 7 months for both study periods.
  Changes from baseline in glucocorticoid dose expressed in prednisone equivalents (mg/day) will be assessed as a measure of steroid tapering over time.
Total Improvement Score (TIS) improvement category (minimal, moderate, or major improvement) in the 2016 ACR/EULAR Myositis Response Criteria | From baseline to 7 months for both study periods.
  Response relative to baseline will be assessed in terms of Total improvement category (minimal TIS ≥20, moderate TIS ≥40, or major TIS ≥60). TIS is a weighted average of the sub-scores in the 6 core set measures that comprise the validated outcome measure in the 2016 ACR/EULAR Myositis Response Criteria.
Total Improvement Score (TIS, expressed as continuous variable) in the 2016 ACR/EULAR Myositis Response Criteria after each repeat dose | From baseline to 1 month, 4 months, and 7 months for both study periods.
  Response to repeat dosing will be assessed by TIS (scale of 0 to 100 points) at 1 month after each repeat dose: TIS at 1 month (after 1 dose), 4 months (after 2 doses), and 7 months (after 3 doses).
Modified Cutaneous Dermatomyositis Disease Area and Severity Index (CDASI) Activity Score | From baseline to 7 months for both study periods.
  The mean changes in the modified CDASI activity score (scale of 0-100) will be assessed. The CDASI is a partially validated, clinician-scored, 1-page outcome measure for assessing skin disease in DM patients. It evaluates the skin in 15 anatomic locations and provides two separate scores based on activity and damage. The CDASI activity score reflects the presence and severity of active skin inflammation, and it is the sum of scores for erythema, scaling, ulceration/erosion, and activity due to Gottron's papules on the hands, recent hair loss, and periungual changes. Higher scores indicate greater disease severity.
Modified Cutaneous Dermatomyositis Disease Area and Severity Index (CDASI) Damage Score | From baseline to 7 months for both study periods.
  The mean changes in the modified CDASI damage score (scale of 0-32) will be assessed. The CDASI is a partially validated, clinician-scored, 1-page outcome measure for assessing skin disease in DM patients. It evaluates the skin in 15 anatomic locations and is comprised of two separate scores based on activity and damage. The CDASI damage score reflects the chronic manifestations of skin disease, and it is the sum of scores for poikiloderma and calcinosis and damage due to Gottron's papules on the hands, recent hair loss, and periungual changes. Higher scores indicate greater disease severity.
Myositis Disease Activity Assessment Tool (MDAAT) | From baseline to 7 months for both study periods.
  The mean changes in scores on the MDAAT will be assessed. The MDAAT utilizes Visual Analogue Scale (VAS). The VAS is a 10-point scale (left end of line = no evidence of disease activity, midpoint of line = moderate disease activity, and right end of line = extreme or maximum disease activity) which the physician assesses, for each of several pre-designated extra-muscular organ systems. The common format is a horizontal bar or line. Physicians assess each designated organ system based on how active the patient's disease has been within the prior four weeks. These VAS ratings are determined with the help of a listed set of clinical and laboratory findings.
Myositis Damage Index (MDI) Extent Score | From baseline to 7 months for both study periods.
  The mean changes in scores on the myositis damage index (MDI) extent score will be assessed. Each organ system is scored 0 or 1 (0 means never present and 1 means present for at least 6 months). The total extent score is the sum of all items scored across all systems divided by the total possible maximum score (scale of 0 to 38 in adults).
Myositis Damage Index (MDI) Severity Score | From baseline to 7 months for both study periods.
  The mean changes in scores on the myositis damage index (MDI) Severity Score will be assessed. Clinician rates the severity of the damage of each organ system using a 10 cm visual analogue scale (VAS) from 0 to 10 (0 means no damage and 10 means extreme damage). Final score is the sum of all systems (scale of 0 to 110 for all 11 systems).
Cutaneous Dermatomyositis Investigator Global Assessment (CDM-IGA) | From baseline to 7 months for both study periods.
  The mean changes in scores on the CDM-IGA will be assessed. The CDM-IGA observes the skin on 11 areas of the body, which are scored on a scale of 0 to 4 based on color and extent of the active cutaneous disease. The final CDM-IGA score is equal to the highest scoring characteristic.
Self-reported physical function capability measured by PROMIS PF-20a | From baseline to 7 months for both study periods.
  The mean change in self-reported physical function capability in each treatment group as measured by PROMIS PF-20 will be assessed. The PROMIS PF-20 measures asks 20 questions about the functioning of the upper extremities (dexterity), lower extremities (walking or mobility), and central regions (neck, back), as well as instrumental activities of daily living, such as running errands. The PROMIS PF-20a provides a single Physical Function capability score and assesses current function.
Glucocorticoid Dose (prednisone equivalents per day) Tapering after repeat doses of study treatment | Baseline, from 3 months to 4 months, and from 6 months to 7 months, for each study period.
  The mean change from baseline in glucocorticoid dose expressed in prednisone equivalents (mg/day) will be assessed as a measure of steroid tapering after two and three doses of study treatment.
Time to achieve maximum TIS improvement category | From baseline to within 7 months for each study period.
  The time (months) from study treatment initiation to when the maximum improvement category is achieved in TIS will be assessed. The improvement in each subject will be categorized as minimal (≤ 20 points change), moderate (21 - 40 points), or major (> 40 points).
Time to confirmed deterioration in the TIS expressed as continuous variable | From baseline to each visit within 7 months for each study period.
  The time (months) from study treatment initiation to confirmed deterioration in TIS (continuous variable, scale of 0 to100) will be assessed.
Pulmonary function test - Forced Expiratory Volume in one second (FEV1) | From baseline to 7 months for both study periods.
  Pulmonary function will be evaluated for normal or abnormal based on the Forced Expiratory Volume in one second (FEV1, Liters) measured by spirometry. FEV1 measures how quickly air can be exhaled in the first second of a forced exhalation. A low FEV1 indicates difficulty with quick air flow out of the lungs, such as in obstructive lung disease. Changes will be assessed.
Pulmonary function test - Forced Vital Capacity (FVC) | From baseline to 7 months for both study periods.
  Pulmonary function will be evaluated for normal or abnormal based on the Forced Vital Capacity (FVC, Liters) measured by spirometry. FVC measures the maximum amount of air a person can forcefully blow out after taking the deepest possible breath. A low FVC can result from poor effort or conditions that restrict the ability of the lungs to fill, such as in restrictive lung diseases. Changes will be assessed.
Pulmonary function test - FEV1/FVC ratio | From baseline to 7 months for both study periods.
  Pulmonary function will be evaluated for normal or abnormal based on the ratio of spirometry measurements of FEV1/FVC (%). The FEV1/FVC ratio helps differentiate between obstructive lung diseases (like asthma or COPD, which lead to disproportionately low FEV1) that result in low FEV1/FVC ratio, and restrictive lung diseases (like pulmonary fibrosis, which lead to low FVC) that can have FEV1/FVC ratio appear normal or high. Changes will be assessed.
Pulmonary function test - Peak Expiratory Flow (PEF) | From baseline to 7 months for both study periods.
  Pulmonary function will be evaluated for normal or abnormal based on the Peak Expiratory Flow (PEF, Liters per second) measured by spirometry. PEF measures the maximum speed (flow rate) at which air can be exhaled from the lungs after a deep breath. A high PEF indicates strong lung airflow, and a low PEF suggests potential issues like airway obstruction. Changes will be assessed.
Pulmonary function test - Diffusing Capacity of the Lungs for carbon monoxide (DLCO) | From baseline to 7 months for both study periods.
  Pulmonary function will be evaluated for normal or abnormal based on the Diffusing Capacity of the Lungs for Carbon monoxide (DLCO, %). DLCO measures the efficiency of gas exchange in the lungs. A normal DLCO indicates healthy gas exchange in the lungs. A low DLCO may suggest possible reduction in the surface area for gas exchange or possible issue with blood flow or blood vessels in the lungs. DLCO is typically measured along with other pulmonary function tests, such as spirometry. Changes will be assessed.
Left ventricular function evaluated by transthoracic echocardiography | From baseline to 7 months for both study periods.
  Left ventricular function will be evaluated for normal or abnormal based on transthoracic echocardiography (TTE) parameters measuring left ventricular ejection fraction (LVEF), left ventricular end diastolic volume (LVEDV), and left ventricular end systolic volume (LVESV).
Functional Index-3 (FI-3) test | From baseline to 7 months for both study periods.
  Changes in endurance of repetitive muscle activity will be assessed by the Functional Index-3 (FI-3) test. The FI-3 is a validated method for assessing functional disability (i.e., muscle endurance and stamina) in patients with DM or PM. The assessment consists of 3 tasks, performed either unilaterally or bilaterally, to test shoulder, neck, and hip flexion, with a total score (0-100) computed from the task results. For this study, neck (30), arm (60), and leg lifts (60) on dominant side will be tested using metronome.
Myositis Antibody Panel | From baseline to 7 months for both study periods.
  Changes in disease activity will be assessed using the extended myositis specific antibody panel IgG titers as biomarkers of myositis disease activity.

OTHER OUTCOMES:
Erythrocyte Sedimentation Rate (ESR) - systemic inflammatory/immune marker | From baseline to 7 months for both study periods and post-study follow-up at 25 months.
  Changes in erythrocyte sedimentation rate (ESR, mm/hour) will be measured as a systemic inflammatory/immune marker. The ESR lab test measures the rate at which red blood cells (erythrocytes) settle in a vertical blood tube over one hour. During inflammation, blood proteins increase that result in ESR increase.
C-Reactive Protein (CRP) - systemic inflammatory/immune marker | From baseline to 7 months for both study periods and post-study follow-up at 25 months.
  Changes in C-Reactive Protein (CRP, mg/L) will be measured as a systemic inflammatory/immune marker in serum samples using a high-sensitivity CRP (HS-CRP) imunoturbidimetric test.
TGF-β1 - systemic inflammatory/immune marker | From baseline to 7 months for both study periods and post-study follow-up at 25 months.
  Changes in cytokine levels of transforming growth factor-beta 1 (TGF-β1, pg/mL) will be measured as a systemic inflammatory/immune marker in plasma samples using a Luminex-based assay panel.
TNF-α - systemic inflammatory/immune marker | From baseline to 7 months for both study periods and post-study follow-up at 25 months.
  Changes in cytokine levels of tumor necrosis factor-alpha (TNF-α, pg/mL) will be measured as a systemic inflammatory/immune marker in plasma samples using a Luminex-based assay panel.
IL-1β - systemic inflammatory/immune marker | From baseline to 7 months for both study periods and post-study follow-up at 25 months.
  Changes in cytokine levels of interleukin-1 beta (IL-1β, pg/mL) will be measured as a systemic inflammatory/immune marker in plasma samples using a Luminex-based assay panel.
IL-1ra - systemic inflammatory/immune marker | From baseline to 7 months for both study periods and post-study follow-up at 25 months.
  Changes in cytokine levels of interleukin-1 receptor antagonist (IL-1ra, pg/mL) will be measured as a systemic inflammatory/immune marker in plasma samples using a Luminex-based assay panel.
IL-2 - systemic inflammatory/immune marker | From baseline to 7 months for both study periods and post-study follow-up at 25 months.
  Changes in cytokine levels of interleukin-2 (IL-2, pg/mL) will be measured as a systemic inflammatory/immune marker in plasma samples using a Luminex-based assay panel.
IL-4 - systemic inflammatory/immune marker | From baseline to 7 months for both study periods and post-study follow-up at 25 months.
  Changes in cytokine levels of interleukin-4 (IL-4, pg/mL) will be measured as a systemic inflammatory/immune marker in plasma samples using a Luminex-based assay panel.
IL-6 - systemic inflammatory/immune marker | From baseline to 7 months for both study periods and post-study follow-up at 25 months.
  Change in cytokine levels of interleukin-6 (IL-6, pg/mL) will be measured as a systemic inflammatory/immune marker in plasma samples using a Luminex-based assay panel.
IL-8 - systemic inflammatory/immune marker | From baseline to 7 months for both study periods and post-study follow-up at 25 months.
  Changes in cytokine levels of interleukin-8 (IL-8, pg/mL) will be measured as a systemic inflammatory/immune marker in plasma samples using a Luminex-based assay panel.
IL-10 - systemic inflammatory/immune marker | From baseline to 7 months for both study periods and post-study follow-up at 25 months.
  Changes in cytokine levels of interleukin-10 (IL-10, pg/mL) will be measured as a systemic inflammatory/immune marker in plasma samples using a Luminex-based assay panel.
IL-17A - systemic inflammatory/immune marker | From baseline to 7 months for both study periods and post-study follow-up at 25 months.
  Changes in cytokine levels of interleukin-17A (IL-17A, pg/mL) will be measured as a systemic inflammatory/immune marker in plasma samples using a Luminex-based assay panel.
IFN-γ - systemic inflammatory/immune marker | From baseline to 7 months for both study periods and post-study follow-up at 25 months.
  Changes in cytokine levels of interferon gamma (IFN-γ, pg/mL) will be measured as a systemic inflammatory/immune marker in plasma samples using a Luminex-based assay panel.
IP-10/ CXCL10 - systemic inflammatory/immune marker | From baseline to 7 months for both study periods and post-study follow-up at 25 months.
  Changes in chemokine levels of interferon gamma-induced protein 10 (IP-10/ CXCL10, pg/mL) will be measured as a systemic inflammatory/immune marker in plasma samples using a Luminex-based assay panel.
Leukocyte phenotyping (if feasible) | From baseline to 7 months for both study periods and post-study follow-up at 25 months.
  Changes in leukocyte, lymphocyte effector, and regulatory phenotype profiles will be assessed by flow cytometry analysis of CD3+, CD4+, and CD8+; CD25+/Foxp3+ cells.
Monocyte M1 and M2 phenotyping (if feasible) | From baseline to 7 months for both study periods and post-study follow-up at 25 months.
  Changes in Monocyte M1 and M2 phenotyping (CD14+, CD16+, CD200+) will be assessed by flow cytometry analysis.
PROMIS Fatigue 13a (FACIT Fatigue Scale) | From baseline to 7 months for both study periods and post-study follow-up at 25 months.
  Changes in patient responses on the PROMIS Fatigue 13a (FACIT Fatigue Scale) questionnaire will be evaluated. This is a 13-item measure that assesses self-reported fatigue and its impact upon daily activities and function during the past week. The level of fatigue is measured on a four point Likert scale (4 = not at all fatigued to 0 = very much fatigued), and the Score is the sum of the scores for all 13 items. The Score range is from 0 to 52; a score of less than 30 indicates severe fatigue, and higher scores indicate better quality of life.
Patient Global Assessment of Pain (PtGA-Pain) | From baseline to 7 months for both study periods and post-study follow-up at 25 months.
  Changes in patient responses on the Patient Global Assessment of Pain (PtGA-Pain) will be evaluated. The PtGA-Pain is a tool for recording patient reported pain levels without use of Visual Analog Scale (VAS).
Physician Global Disease Activity Visual Analog Scale (VAS) - TIS Core Set Measure 1 of 6 | From baseline to 7 months for both study periods and post-study follow-up at 25 months.
  Changes in the Physician Global Disease Activity Visual Analog Scale (VAS) TIS sub-score will be assessed. The VAS is a 10-point scale, across which a respondent selects a point that best reflects the intensity of disease activity. The common format is a horizontal bar or line. The VAS is anchored at each end by terms that describe disease severity extremes: 0 for no disease activity, and 10 for the most severe disease activity. The IIM six core set measures include three VAS 10 scales, consisting of physician-reported, patient-reported, and extramuscular disease activity.
Patient Global Disease Activity (VAS) - TIS Core Set Measure 2 of 6 | From baseline to 7 months for both study periods and post-study follow-up at 25 months.
  Changes in the Patient Global Disease Activity (VAS) TIS sub-score will be assessed. The VAS is a 10-point scale, across which a respondent selects a point that best reflects the intensity of disease activity. The common format is a horizontal bar or line. The VAS is anchored at each end by terms that describe disease severity extremes: 0 for no disease activity, and 10 for the most severe disease activity. The IIM six core set measures include three VAS 10 scales, consisting of physician-reported, patient-reported, and extramuscular disease activity.
Manual Muscle Strength Test (MMT-8) - TIS Core Set Measure 3 of 6 | From baseline to 7 months for both study periods and post-study follow-up at 25 months.
  Changes in the MMT-8 TIS sub-score will be assessed. The MMT-8 testing is performed as part of the 2016 ACR/EULAR Myositis Response Criteria for Minimal, Moderate, and Major Clinical Response in Adult Dermatomyositis and Polymyositis and is a series of physical tasks done by the patient in tandem with the physician to assess resistance and endurance on target muscles (some of which overlap with the FI-3 below) for an overall score between 0 and 80 (when assessed unilaterally).
Health Assessment Questionnaire Disability Index (HAQ-DI) - TIS Core Set Measure 4 of 6 | From baseline to 7 months for both study periods and post-study follow-up at 25 months.
  Changes in the HAQ-DI TIS sub-score will be assessed. The HAQ was developed as a comprehensive measure of outcome in patients with a wide variety of rheumatic diseases. There are 8 sections: dressing, arising, eating, walking, hygiene, reach, grip, and activities. There are 2 or 3 questions for each section. Scoring within each section is from 0 (without any difficulty) to 3 (unable to do). For each section the score given to that section is the worst score within the section, i.e. if one question is scored 1 and another 2, then the score for the section is 2. In addition, if an aid or device is used or if help is required from another individual, then the minimum score for that section is 2. If the section score is already 2 or more then no modification is made.
Extramuscular Disease Activity (VAS) - TIS Core Set Measure 5 of 6 | From baseline to 7 months for both study periods and post-study follow-up at 25 months.
  Changes in the Extramuscular Disease Activity (VAS) TIS sub-score will be assessed. The VAS is a 10-point scale, across which a respondent selects a point that best reflects the extramuscular disease activity. The common format is a horizontal bar or line. The VAS is anchored at each end by terms that describe disease severity extremes: 0 for no disease activity, and 10 for the most severe disease activity. The IIM six core set measures include three VAS 10 scales, consisting of physician-reported, patient-reported, and extramuscular disease activity.
Muscle Enzymes - TIS Core Set Measure 6 of 6 | From baseline to 7 months for both study periods and post-study follow-up at 25 months.
  Changes in the TIS sub-score for serum level of muscle enzymes will be assessed.
The percentage of patients by treatment group who met the criteria for clinical deterioration | From baseline to within 7 months for each study period.
  The percentage of participants in each cohort who met the criteria for clinical deterioration up to 7 months will be assessed.
The percentage of participants in each cohort who require rescue therapy other than steroids | From baseline to within 7 months for each study period.
  The percentage of participants in each cohort who require rescue therapy other than steroids will be assessed.

CONTACTS AND LOCATIONS:
Overall Officials: Michael Bubb, MD, Principal Investigator — Malcom Randall North Florida/South Georgia VA Medical Center
Locations (2):
- United States (2):
  - Malcom Randall North Florida/South Georgia VA Medical Center, Gainesville, Florida
  - Bioresearch Partner, Miami, Florida